CLINICAL TRIAL: NCT05702320
Title: Investigation of the Effect of Reflective Blanket on Reducing the Development of Undesirable Perioperative Hypothermia
Brief Title: Effect of Reflective Blanket on Undesirable Perioperative Hypothermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Öğr. Gör. Ali GÜZEL (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Sponsor-Investigator, Öğr. Gör. Ali GÜZEL, principal investigator, Bitlis Eren University
Organization: Bitlis Eren University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2021/041
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Abdominal Surgery; General Anesthesia; General Surgery
Keywords: unwanted perioperative hypothermia; reflective blanket; general anesthesia; Abdominal surgery

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental research
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reference Group (Experimental): Patients in this group will be warmed for 15 minutes with a full-body blanket belonging to the air-blown heater device before surgery. The heating will be Decelerated until he is taken to the operating table, and after the preparations are completed, the lower extremities will continue to be heated with a half-body blanket belonging to the heating device. After the patient is taken to the post-anesthesia care unit, the soaked blankets will be removed and the whole body will continue to be warmed with a blanket as in the preoperative period. When the patient's body temperature rises above 36 °C, the heating process will be terminated and when he meets the criteria for being transferred to the clinic, his transfer to the clinic will be provided in accordance with the institution's policy.
  Interventions: Other: the heating procedure
- intervention group (Experimental): The patients in this group will be wrapped with a reflective blanket from the neck to the whole body with the reflective side facing the patient for 15 minutes before the operation, so that only the surgical gown is on the patients in this group. After a layer of operating room cover is placed on the patient's lower extremities on the operating table in accordance with the hospital procedure, a reflective blanket will be wrapped on it with the reflective side facing the patient. After the patient is taken to the post-anesthesia care unit, the soaked covers will be removed and the entire body of the patient will be wrapped with a reflective blanket, as in the preoperative period. When the patient's body temperature rises above 36 °C and he meets the criteria for being transferred to the clinic, his transfer to the clinic will be provided in accordance with the institution's policy.
  Interventions: Other: the heating procedure
- control group (No Intervention): No heating procedure will be performed by the researcher in this group of patients during the perioperative period, only the number of covers provided for heating in the post-anesthesia care unit will be recorded. The duration of stay in the post-anesthesia care unit, the transfer of the patient to the clinic and the follow-up in the clinic will be carried out according to the hospital procedure.

INTERVENTIONS:
Other: the heating procedure — The patients will undergo a heating procedure.
  Arms: Reference Group; intervention group

SUMMARY:
The aim of this study is to determine the effect of using reflective blankets, which is a passive insulation product, on preventing UPH in patients scheduled for abdominal surgery under general anesthesia. It will also be evaluated whether the reflective blanket has an effect on the patients' thermal comfort and shivering levels. Inconsistent results have been reported in studies using reflective blankets. This inconsistency may be due to the fact that it was used at different stages of the perioperative process or that the body was not adequately isolated. In this study, we aimed to use the reflective blanket throughout the perioperative process and to isolate the patient's body as much as possible. Reflective blankets are inexpensive, practical to use and easy to store. With the positive results that can be obtained from this study, it can be used not only in operating rooms, but also in intensive care or other services where hypothermia is likely to occur.

Within the scope of the study, a Reference group (warm air blower device), an Intervention group (reflective blanket) and a Control group (routine hospital procedure) will be established. The study was planned to be conducted with a total of 102 patients, with 34 patients in each group.

In this study; patients' vital signs, coagulation tests, thermal comfort and shivering levels will be evaluated. Patients in the Reference and Intervention group will be warmed before the surgery (15 minutes), during the surgery, and until they are transferred from the post-anaesthetic care unit to the clinic. No heating process will be applied to the control group by the researcher. All patients transferred to the clinic will undergo the routine care procedure of the hospital.

DETAILED DESCRIPTION:
Undesirable perioperative hypothermia (UPH) is a decrease in the core body temperature, expressed as the temperature of the blood and internal organs, below 36°C. UPH is an important complication of -anesthesia- and surgery and can occur during the period from the preoperative period (1 hour before anesthesia) to the postoperative period (the first 24 hours after anesthesia). There is a risk of developing UPH in all patients who will undergo surgery.

The application of general anesthesia, the cold environment of the operating room, the openness of the operated internal body region to ambient temperature, the long duration of the operation, the use of unheated IV fluids and irrigation fluids contribute to the development of UPH. Body temperature loss occurs rapidly with four mechanisms in the form of radiation, conduction, convection and evaporation before anesthesia and after anesthesia induction.

UPH causes many undesirable negative consequences for the patient. The deterioration of these patient comfort, flicker, myocardial problems, wound infection, wound healing problems, postoperative pain, platelet dysfunction, increased blood loss and blood transfusion requirements, renal function deterioration, a decrease in drug metabolism, anesthesia, post-operative care unit and prolong the length of stay in hospital and is expressed in the increase of mortality.

In the perioperative process, two methods are used to warm patients in the form of active and passive heating (insulation). Active heating, hot air blown systems, electric drapes (resistive systems), radiant heaters, intravenous fluids, blood, blood-product heaters, heat and moisture exchanger, filters, heating methods include negative pressure. While systems with hot air blowing reduce heat loss by radiation, they also provide temperature increase by convection. Heating devices should be used together with special suitable blankets and these blankets should cover as much of the body as possible. Cotton-wool blankets, socks, surgical drapes or plastic drapes with metal additives are used for passive heating. The effect of passive insulation is directly proportional to the area covered. Passive heating is recommended to prevent hypothermia in patients with a body temperature of 36 °C and above, and active heating is recommended in patients with a body temperature of less than 36°C.

It is stated that patients who are scheduled for general anesthesia should be warmed up for at least 10-20 minutes before surgery.The combination of more than one heating technique to ensure normothermia increases the effectiveness. Heating with hot air blowing devices is a widespread and effective approach to achieving normothermia and patient satisfaction. The superiority of these devices has been proven in many studies. On the other hand, providing a heating unit for each patient both in the operating room and in the post-anesthesia care unit will cause a serious cost increase.

Interest in passive insulation products has increased due to the cost of hot air blown devices. Passive heating covers that reflect radiant body heat to prevent excessive heat loss to the cold operating room environment can be an alternative to hot air blown devices. The use of such covers does not affect the laminar airflow and eliminates the transfer of potentially pathogenic organisms, since they do not have reusable parts. One of these passive insulation products is reflective blankets. Reflective blankets; it is also referred to by different names such as space blanket, burn blanket, shock blanket and emergency blanket. Reflective blankets were introduced in the 1960s and were originally used for survival purposes. In particular, they contain a metallized plastic layer that reduces heat loss due to radiation and convection. They do not give off heat from the outside, they function by reflecting the heat emitted from the body. It has been reported that reflective blankets reflect 80% of the emitted body heat and can reduce radiant heat loss from 100 kcal to 40 kcal per hour.

Inconsistent results have been reported in studies using reflective blankets. This discrepancy may be due to the fact that it has been used at different stages of the perioperative process or that the body has not been sufficiently isolated.

Purpose and objectives:

The aim of the research is to determine the effect of using a reflective blanket, which is a passive insulation product, on the prevention of UPH in patients who are scheduled for abdominal surgery under general anesthesia. At the same time, it will also be evaluated whether the reflective blanket has an effect on the thermal comfort and shivering levels of the patients.

In line with the current goal, it is planned to achieve the following goals. Goal 1: To ensure that the current body temperature of the patients to be operated is maintained.

Goal 2: To prevent the development of UPH in patients undergoing surgery. Goal 3: To prevent trembling and to ensure thermal comfort in operated patients.

With the positive results that can be obtained from the research; recommendations accompanied by scientific evidence will be presented in the direction of preventing hypothermia before it occurs, maintaining normothermy, and increasing patient comfort by preventing chills and chills that are uncomfortable for patients.

METHOD:

The prescribed research period:

12 months

Where the Research Will Be Conducted:

It is planned that the research will be conducted in the operating room and General Surgery clinic of Bitlis State Hospital affiliated to Bitlis Provincial Health Directorate.

The Ethical Aspect of the Research:

* The ethics committee permission was obtained from the Hasan Kalyoncu University Ethics Committee Presidency for the research (Decision no: 2021/041, Decision date 06.12.2021).
* Application permission was obtained from Bitlis Provincial Health Directorate and Bitlis State Hospital for the research (18/02/2022 13:58- E75384813-000-864).

The universe of research:

In the operating room of Bitlis State Hospital, patients who underwent abdominal surgery under general anesthesia during the research process will form.

Sample of the research:

The data of the Randomized controlled trial titled 'Evaluation of Warming Efficacy on Physiological Indices of Patients Undergoing Laparoscopic Cholecystectomy Surgery: A Randomized Controlled Clinical Trial' were used to calculate the sample size of the study due to the similarity of the study design. Within the scope of the study, a Reference group (hot air blowing device), an Intervention group (reflective blanket) and a Control group (routine hospital procedure) will be formed. Power analysis was performed with G*Power for the number of samples of the study, which is in the experimental/control pattern structure. In the study, the effect level of power analysis was taken as 0.25; α value was taken as 0.05 and power value (1- β) was taken as 0.80 and the number of samples was calculated as 102 in total. Accordingly, it is planned to conduct the study with a total of 102 patients, with 34 patients in each group. The research will be continued until the data of at least 34 patients in each group are completed.

Scope and limitations:

In this study; body temperature, arterial blood pressure, pulse, respiration, oxygen saturation, coagulation tests, thermal comfort and tremor levels of the patients will be evaluated. Coagulation tests will be taken from routine test results, no samples will be taken from patients for this study. Since there is no separate unit in the institution where the research will be conducted, preoperative preparations will be made in the post-anesthesia care unit. The temperature and humidity levels in the patient room, operating room room and post-anesthesia care unit will be adjusted according to the institution's policy and measured for each patient during the research process. The patients who are in the 'control group' and 'Intervention group' will be given additional operating room covers in the post-anesthesia care unit if they request October and this situation will be recorded.

The research was conducted during the preoperative period (one hour before the induction of anesthesia), intraoperative period and postoperative period (after anesthesia 24. it will be carried out in three stages (up to one hour). Before starting the research, nurses in the clinic and nurses and anesthesia technicians in the operating room will be informed about the purpose and method of the research and their training will be provided.

In the clinic; patients who meet the sample selection criteria will be informed about the study orally and in writing and invited to participate in the study. For this purpose, a separate form (Volunteer Information and Consent Form) will be prepared by the researcher and patients who agree to participate in the study will be asked to sign it.

Randomization:

Patients who are accepted to participate in the study will be randomly assigned to the 'Reference', 'Intervention' and 'Control' groups according to the types of A, B and C cards contained in the envelope using the closed envelope technique. Thus, those who choose the A card will be taken to the 'Reference' group, those who choose the B card will be taken to the 'Intervention' group, and those who choose the C card will be taken to the 'Control' group. The randomization process will be created by an impartial medical staff who is not involved in the research. Whichever group the patient is assigned to, oral and visual information will be given about the heating procedures to be applied within the scope of the research.

Data collection tools and data collection:

In the study, patients with identifiable information, vital signs (body temperature, arterial blood pressure, pulse, respiration, oxygen saturation), coagulation tests, and flicker levels of thermal comfort data will be obtained. For this purpose, the forms evaluating the thermal comfort and tremor levels and the follow-up charts prepared by the researcher will be used. Body temperature will be monitored through the tympanic membrane due to the advantage of use in the entire perioperative process, taking into account the recommendations of the guidelines. The tympanic thermometer to be used for measuring body temperature will be calibrated according to the institution's policy. A pulse oximeter device will be used for pulse and oxygen saturation measurements before the patient enters the operating room and in the clinic after surgery, and a patient head monitor will be used at other stages. Arterial blood pressure data will be obtained manually in the clinic before the patient enters the operating room and after surgery, and at other stages with a bedside monitor. Respiratory count data will be obtained by using a second clock in the clinic before the patient enters the operating room and after surgery, and at other stages by a bedside monitor. A patient head monitor belonging to the hospital will be used in the research. For arterial blood pressure measurement, the ERKA brand Perfect Aneroid Model Adult Blood Pressure Monitor (Germany), which was provided by the responsible researcher, will be used.

Identifying data of the patient:

Before the surgery, the study group prepared by the researcher in line with the literature and in which the patients were taken will be recorded through a form containing information such as gender, age, height, weight, body mass index (BMI), chronic disease, if any, the surgical procedure performed, ASA score and fasting time before surgery.

Thermal Comfort Perception Assessment Form:

By the researcher, in line with the literature was prepared. According to the form: 0 refers to extremely unbearable cold, 50 is the ideal temperature (neither hot nor cold), and 100 refers to extremely unbearable temperature. Patients will be asked to mark the place expressing their immediate condition.

Tremor Level Assessment Form:

This form, which was used to evaluate the patient's tremor level, was prepared in accordance with the literature. The level of tremor will be evaluated based on observation in the form of 0 (absent), 1 (mild; tremor localized only in the neck and / or thorax), 2 (moderate; tremor in the neck, upper extremities of the thorax) and 3 (severe; tremor in the trunk, upper and lower extremities).

Defining Points 0 No tremors

1. Mild: Tremor localized only in the neck and/or thorax
2. Moderate: Tremor in the neck, thorax upper extremities,
3. Severe: Tremor in the trunk, upper and lower extremities,

The Heating Procedure:

In order for preoperative heating to be applied, patients with a 'Reference group' and an 'Intervention group' will be taken to the waiting unit at least 20 minutes before the operation. Patients in the control group will be taken from the clinic to the operating room according to the hospital procedure.

1. Reference group:

   Active heating of patients is considered the gold standard for the prevention of UPH and maintenance of normothermy. In this research, it is one of the active heating methods and its superiority has been proven in many studies the heating procedure with hot air blowing devices will be followed as a 'Reference group'. Patients in this group will be taken from the clinic to the preoperative waiting unit wearing surgical gowns. Patients will be covered from the neck up with a full body blanket belonging to the warm air blown heater device before the operation, so that only the surgical gown is on, and the temperature setting will be selected according to the manufacturer's recommendation. The heating time will be 15 minutes. The heating will be Decelerated until he is taken to the operating table, and after the preparations are completed, the lower extremities will continue to be heated with a half-body blanket belonging to the heating device. When the body temperature rises above 37°C, the heating process will be terminated. Sterile covers can be covered on the heating blanket in accordance with the institution's policy. After the patient is taken to the post-anesthesia care unit, the soaked blankets will be removed and the whole body will continue to be warmed with a blanket as in the preoperative period. When the patient's body temperature rises above 36 °C, the heating process will be terminated, and when he meets the criteria for being transferred to the clinic, his transfer to the clinic will be provided in accordance with the institution's policy. After this stage, the standard heating procedure of the hospital will be applied to the patients.
2. Intervention group:

   Patients in this group will be taken from the clinic to the preoperative waiting unit wearing surgical gowns. The patients will be wrapped with a reflective blanket from the neck to the whole body with the reflective side facing the patient for 15 minutes before the operation, so that only the surgical gown is on the patients. The blanket will remain wrapped until he is taken to the operating table. After a layer of operating room cover is placed on the patient's lower extremities on the operating table in accordance with the hospital procedure, a reflective blanket will be wrapped on it with the reflective side facing the patient. Sterile covers will be covered on the reflective blanket in accordance with the institution's policy. After the patient is taken to the post-anesthesia care unit, the soaked covers will be removed and the entire body of the patient will be wrapped with a reflective blanket, as in the preoperative period. If the patient requests, he will October be covered with operating room covers and this situation will be recorded. When the patient's body temperature rises above 36°C and he meets the criteria for being transferred to the clinic, his transfer to the clinic will be provided in accordance with the institution's policy. After this stage, the standard heating procedure of the hospital will be applied to the patients.
3. Control group:

The standard heating procedure of the hospital will be applied to the patients in this group. In this standard procedure, patients are taken to the operating room shortly before the operation by removing all their clothes in the clinic and wearing only an operating room apron. Patients are taken directly to the operating room without waiting, except for unexpected delays in the operating room, the operating room is not ready at that time, etc. No heating procedure is applied to the patients in this group during the preoperative period, and passive heating is provided with the covers belonging to the operating room in the intraoperative process and post-anesthesia care unit. No heating procedure will be performed by the researcher in this group of patients during the perioperative period, only the number of covers provided for heating in the post-anesthesia care unit will be recorded. The duration of stay in the post-anesthesia care unit, the transfer of the patient to the clinic and the follow-up in the clinic will be carried out according to the hospital procedure.

Obtaining data of the preoperative period:

While wearing the surgical gown in the clinic, the data of body temperature, arterial blood pressure, pulse, respiration, oxygen saturation, thermal comfort and tremor levels of all patients will be taken. The patients in the 'Reference' and 'Intervention' groups will be taken to the waiting unit 15 minutes before the operation, enough time for the heating procedure to be performed. The control group patients will be followed according to the hospital procedure. Data for this period; the time of leaving the patient's room, the temperature, humidity of the patient's room, the time of admission to the waiting unit, the temperature, humidity of the unit, etc. will be recorded through a form prepared by the researcher containing the characteristics and vital signs. 'Reference' and 'Intervention' in the group of patients with Tremor and other vital signs body temperature and thermal comfort levels; at the entrance to the operating room unit, then 15 minutes, and the most recent surgery will be taken before entering the Hall. The data of the control group patients will be taken at the entrance to the operating room unit and immediately before entering the operating room.

Obtaining data of the intraoperative period:

All patients belonging to all three groups will have their body temperature measured tympanically when they are taken to the operating room, and body temperature and other vital signs will continue to be measured at December intervals of 15 minutes from the induction of anesthesia until they are taken to the post-anesthesia care unit. Body temperature will be monitored through the tympanic membrane, and other vital signs will be monitored with a bedside monitor. These findings and the data that belongs to the operating theatre (type of surgery <Laparoscopic/open>, entry time to the operating room, the operating room, temperature/humidity, the time of induction of anesthesia, the operating room from the entrance to the period of induction of anesthesia, duration of operation, termination of anesthesia time, recovery time from anesthesia, after anesthesia care unit transfer time from surgery, intraoperative IV fluids given the amount of heating start time <intervention groups>), prepared by the researcher through the form will be recorded.

Data of the post-anesthesia care unit:

When all patients are taken to the post-anesthesia care unit, their body temperature will be measured tympanically, and other vital signs will be measured with a bedside monitor, and they will continue to be measured at December intervals of 15 minutes until the patient is transferred to the clinic. Data for this period; the time of receipt by the researcher prepared and anaesthesia care unit, duration of transfer of the unit to the clinic clock temperature/humidity unit is provided blankets and additional IV fluid given in the amount of time/number of properties such as vital signs (body temperature, arterial blood pressure, pulse, respiration, oxygen saturation) will be recorded through a form that contains. Simultaneously with these data, thermal comfort and tremor levels will also be evaluated. The transfer of the control group patients to the clinic will be made according to the hospital procedure and their findings will be recorded at the time of their transfer to the clinic.

Data of the clinic:

After this stage, all patients will be treated with the standard heating procedure of the hospital. The data for this period will be recorded through a form prepared by the researcher containing information such as the patient's time of admission to the clinic, the patient's room temperature / humidity, vital signs, chills and thermal comfort level. When the patients are taken to the bed (0. data related to body temperature, arterial blood pressure, pulse, respiration, oxygen saturation, thermal comfort and tremor levels will be recorded. Body temperature and oxygen saturation during the first hour (every 15 minutes), the second hour (every 30 minutes) and 4-8 and 24. it will be measured in hours. Arterial blood pressure, pulse and respiratory rate, after admission to the sickbed, 0-60-90-120. in minutes and 4-8-12 and 24. it will be measured in hours. Thermal comfort 0-30-60-90-120. minutes and 4 and 8. it will be evaluated within hours. The tremor levels are 0-15-30-45-60-90 and 120. it will be evaluated in minutes.

Statistical Analysis of the Data:

In the research, the analysis of the data will be carried out with the SPSS for Windows program and the results will be evaluated at the 95% confidence level. Within the scope of the study, kurtosis and skewness coefficients will be calculated to determine the suitability of quantitative data for normal distribution, and Kolmogrow-Simirnow tests will be examined. However, ANOVA test will be performed when comparing the three groups, and if there is a significant difference, a double comparison will be made with the post hoc test.

ELIGIBILITY:
Inclusion Criteria:

* abdominal surgery is planned,
* ASA I-II patients,
* who will undergo general anesthesia,
* operations where the anesthesia time is expected to take 30-120 minutes
* the age of 18,
* with a body mass index of 18.5-35 kg/m2,
* who can read and write,
* who participate voluntarily.

Exclusion Criteria:

* Patients who used any corticosteroids or other immunosuppressive drugs four weeks before surgery,
* Patients with a recent history of fever and/or infection,
* Patients with hypopituiterism,
* Patients taking antipsychotics and antidepressants,
* Patients with diabetic neuropathy,
* Active otitis media patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-02-14 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Does the application of passive insulation with a reflective blanket during the perioperative process reduce the incidence of unwanted Perioperative Hypothermia in patients? | 12 months
  Passive heating will be applied with a reflective blanket, body temperatures will be measured and the results will be recorded.
Does the application of passive insulation with a reflective blanket during the perioperative process reduce the incidence of tremors in patients? | 12 months
  Passive heating will be applied with a reflective blanket, the tremor status of the patients will be measured with the tremor level assessment form and the results will be recorded.
Does the application of passive insulation with a reflective blanket during the perioperative period increase the level of thermal comfort perception in patients? | 12 months
  Passive heating will be applied with a reflective cover, the thermal comfort levels of the patients will be measured with a thermal comfort perception assessment form and the results will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No